CLINICAL TRIAL: NCT01246908
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Assessment of the Efficacy, Safety and Tolerability of CX157 Modified Release Tablet, 125 mg Twice Per Day in Subjects With Treatment Resistant Depression
Brief Title: Efficacy, Safety and Tolerability of CX157 in Treatment Resistant Depression
Acronym: CX157-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CeNeRx BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX157-201
Record Dates: First submitted 2010-11-02; First posted 2010-11-24 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Treatment Resistant Depression
Keywords: TRD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Sugars; CX157

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CX157 (TriRima) (Experimental): CX157 (TriRima) in a reversible monoamine oxidase inhibitor (MAOI)
  Interventions: Drug: CX157 (TriRima)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo administered twice per day for six weeks.
  Other Names: Sugar Pill
  Arms: Placebo
Drug: CX157 (TriRima) — One tablet administered twice per day (total daily dose of 250 mg) for six weeks.
  Arms: CX157 (TriRima)

SUMMARY:
The purpose of this study is to determine if CX157 is effective and safe in patients with treatment of treatment resistant depression over six weeks of treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to examine the efficacy of CX157 Modified Release Tablet, 125 mg administered twice per day (BID) as compared to placebo in subjects with Treatment Resistant Depression (TRD). Secondary objectives are to evaluate the safety and tolerability of CX157 Modified Release Tablet, 125 mg BID in TRD subjects and characterize steady-state pharmacokinetic profile and explore pharmacodynamic relationships.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 20 to 65 years of age
2. Able to read, understand and converse in English and provide written, dated informed consent
3. Diagnosed with Major Depressive Disorder (MDD)and Treatment Resistant Depression(TRD)
4. Females on acceptable method of contraception

Exclusion Criteria:

1. Major depressive episode greater than five years
2. A history of a Substance Use Disorder with the exception of nicotine dependence in the past 12 months
3. Obsessive-Compulsive Disorder (OCD), Panic Disorder, Post-traumatic Stress Disorder (PTSD
4. A history of schizophrenia or schizoaffective disorders
5. A history of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within the past five years
6. A history of Antisocial Personality Disorder or Borderline Personality Disorder
7. Recent suicidal behavior and is at risk of such behavior during the course of the study
8. Electroconvulsive therapy (ECT) within the past five years
9. Transcranial Magnetic Stimulation (TMS) for the treatment of the current episode of depression
10. Vagus Nerve Stimulation (VNS) at any time
11. Any psychoactive drugs within one to four weeks prior to the randomization visit depending on the type of drug
12. Significant abnormality on the screening physical examination
13. Significant cardiac abnormalities such as uncontrolled hypertension, recent myocardial infarction, Congestive heart failure (CHF), Angina pectoris
14. A history within the past two years of significant head trauma, surgical procedure involving the brain,degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation
15. A history of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than six months
16. A history of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening
17. Participation in an investigational study in the past one month
18. A positive screening urine test for drugs of abuse
19. Female subject who is pregnant or lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | Over six weeks of study treatment
  The MADRS will be administered by a trained rater at the study site and assess symptoms of depression.

SECONDARY OUTCOMES:
Severity of illness (CGI-S); | Over six weeks of treatment with study drug.
  To measure severity of depression
Global Improvement (CGI-I) | Over six weeks of treatment
  To measure overall improvment.
Hospital Anxiety Depression Rating Scale (HADS) | over six weeks of treatment
  To measure symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Alan Yeo, MD, Principal Investigator — Summitt Research Network - Oregon; Ram Shrivastava, MD, Principal Investigator — Eastside Comprehensive Medical Center; Angelo Sambunaris, M.D., Principal Investigator — Atlanta Institute of Medicine and Research; Bijan Bastani, M.D., Principal Investigator — NorthCoast Clinical Trials; Mary Stedman, M.D., Principal Investigator — Stedman Clinical Trials; Richard Weisler, M.D., Principal Investigator — Richard H. Weisler, M.D. and Associates; Mark Joyce, M.D., Principal Investigator — Clinical Neuroscience Solutions, Inc.; Fares Arguello, MD, Principal Investigator — Radiant Research; Valerie Arnold, MD, Principal Investigator — Clinical Neurosciences Solutions, Inc.; Arif Khan, MD, Principal Investigator — Northwest Clinical Research Center; Irving Kolin, MD, Principal Investigator — Kolin Research Group; Jelena Kunovac, MD, Principal Investigator — Excell Research; Jerry Steiert, MD, Principal Investigator — Summit Research Network (Seattle) LLC; Lorena Wallhauser, MD, Principal Investigator — Patient Priority Clinical Sites, LLC; Mohammed Bari, MD, Principal Investigator — Synergy Clinical Research Center; Prakash Bhatia, MD, Principal Investigator — Synergy Escondido; Michael Downing, MD, Principal Investigator — FutureSearch Trials of Dallas; David Brown, MD, Principal Investigator — Community Clinical Research, Inc.; Rosario Hidalgo, MD, Principal Investigator — University of South Florida College of Medicine Psychiatry Center; Alec Bodkin, MD, Principal Investigator — Mclean Hospital; Russell Pet, MD, Principal Investigator — AccelRx Research; Beal Essink, M.D., Principal Investigator — Oregon Center for Clinical Investigations, Inc; Scott Segal, M.D., Principal Investigator — The Segal Institute of Clinical Research; Jeffrey Simon, M.D., Principal Investigator — Northbrooke Research Center; Charmaine Semeniuk, M.D., Principal Investigator — Pacific Clinical Research; John Prater, M.D., Principal Investigator — Gulfcoast Clinical Research Center; Mark Woyshville, M.D., Principal Investigator — North Star Medical Research LLC; Nathan Shapira, MD, Ph.D, Principal Investigator — Carman Research; Robert Molpus, MD, Principal Investigator — Clinical Neuroscience Solutions, Inc.
Locations (30):
- United States (30):
  - Synergy Escondido, Escondido, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Pacific Clinical Research, Orange, California
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - The Segal Institute of Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - University of South Florida College of Medicine Psychiatry Center, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Kolin Research Group, Winter Park, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Nathan Shapira, MD, Ph.D, Smyrna, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - AccelRx Research, Fall River, Massachusetts
  - Eastside Comprehensive Medical Center, New York, New York
  - Richard H. Weisler, M.D. and Associates, Raleigh, North Carolina
  - NorthCoast Clinical Trials, Inc., Beachwood, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Oregon Center for Clinical Investigations, Inc, Portland, Oregon
  - Summitt Research Network (Oregon), Portland, Oregon
  - Introspect of Buxmont, Ltd, Colmar, Pennsylvania
  - Clinical Neurosciences Solutions, Inc., Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Radiant Research, Murray, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Northbrooke Research Center, Deer Brown, Wisconsin